CLINICAL TRIAL: NCT01853358
Title: Phase I of Infusion of Selected Donor NK Cells After HLA Identical Allogeneic Stem Cell Transplantation Prepared With Reduced Intensity Conditioning - DLI-NK/IPC 2012-003
Brief Title: Phase I of Infusion of Selected Donor NK Cells After Allogeneic Stem Cell Transplantation
Acronym: DLI-NK
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DLI-NK/IPC 2012-003
Record Dates: First submitted 2013-04-04; First posted 2013-05-15 (Estimated); Last update posted 2018-07-12 (Actual); Status verified 2018-07

CONDITIONS: Hematological Malignancy
Keywords: hematological malignancy; stem cell transplantation
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- NK Cell infusion (Experimental): * Cell collection
    o Lymphocytes will be harvest from the original and consenting donor as soon as possible around day 60 post transplantation
  * NK Cell selection
    o Cells will be obtained after double selection: CD3+ depletion followed by CD56+ selection using an european approved device (Miltenyi corporation)
  * NK Cell ex-vivo activation
    o ex-vivo activation: interleukin-2 according to a classical procedure (7 days at 37°C with RPMI clinical grade medium supplemented with 10% of foetal calf serum, 0.5 x 106 cellules / ml, 1000 U/ml d'IL-2 (interleukin, proleukin)
  * NK Cell infusion (60 to 90 days after transplantation)
  Interventions: Biological: NK Cell infusion

INTERVENTIONS:
Biological: NK Cell infusion — * level 1: 1 x 10e6 NK cells /kg;
  * level 2: 5 x 10e6 NK cells /kg;
  * level 3: > 5.10e6 and ≤ 5.10e7 cellules NK/kg

SUMMARY:
The goal of our study will be to determine the clinical and biological safety of infusing immuno-selected NK (Natural Killer) CD3-/CD56+ cells, early after allogeneic transplantation with colony stimulating factor (G-CSF) mobilized peripheral blood stem cells and Reduced Intensity Conditioning (RIC), as a potential substitute to usual "Donor Lymphocyte Infusion" (DLI), that contain the whole range of immune effectors. The trial will include several progressive steps: dose escalation up to a level compatible with the cost-effectiveness potential of the device and clinical situation and recombinant interleukin-2 (r-IL2) activation of selected NK cells in vitro prior to re-infusion.

DETAILED DESCRIPTION:
In the mid 90's, it has been shown that donor lymphocyte infusions (DLI), when given for Chronic Myelocytic Leukemia (CML) that has relapsed after conventional allogeneic stem cell transplantation (SCT), result in a high incidence of durable cytogenetic and molecular remissions. However, regular documented effects are the occurrence of secondary aplasia and/or graft-versus-host disease (GVHD) including the post RIC situation. These effects are related to the high content of cytotoxic T cells in the DLI. Attempts to deplete CD8+ T-cells from DLI have been conducted with promising results but are not totally satisfactory.

More recently the infusion of r-IL2 ex-vivo activated autologous or allogeneic NK-selected cells have been studied and the safety established in patients presenting various malignancies.

Indeed, NK are thoroughly characterized in terms of genotype, phenotype and function. Although a handful of clinical-grade reagents and devices exist that give access to the human NK cell compartment, an immuno-selection device exists that allows for the selection of NK cells from various types of hematopoietic cell collections in view of clinical applications: the process produces CD3-/CD56+ cells in two steps and have been used in the previous experiences.

ELIGIBILITY:
Inclusion Criteria:

1. Patient treated with allogeneic stem cell transplantation

   * Presenting an hematological malignancy with an intermediate, high or very high risk index according to the disease risk index developed by the Dana Farber Cancer Institute
   * Donor: HLA matched related or unrelated (10/10) donor
   * Graft: Peripheral stem cell transplant
   * Reduced Intensity Conditioning as used in the current transplant program: Fludarabine, IV Busulfan and Thymoglobuline
2. Age above 18 and under 70
3. Eastern Cooperative Oncology Group (ECOG) 0-1 or Karnofsky index ≥ 70 %
4. Survival expectation > 6 months
5. Affiliation to social security
6. Signed informed consent from Donor and Patient

Exclusion Criteria:

1. Active grade >= 2 acute GVHD or corticotherapy ≥ 0.5 mg/kg/day at time of NK cell infusion
2. Active infection
3. Psychiatric disorder occurring after transplant
4. Pregnant or breast-feeding women or without contraception

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Estimated)
Dates: Start 2013-04 (Actual); Primary Completion 2018-03-15 (Actual); Study Completion 2018-03-15 (Actual)

PRIMARY OUTCOMES:
Occurence of grade 3-4 toxicity within 30 days of NK cells infusion | day 30
  To establish the safety of donor NK cells infusion after HLA matched allogeneic transplant prepared by RIC.

SECONDARY OUTCOMES:
Number of infused cells population : CD3+, CD56+/CD16+, CD56-/CD16+, CD56+/CD16- (Determination) | baseline: at the time of the NK cells infusion
  Ex vivo NK cell selection reproductibility
relapse | up to one year after infusion
number of NK cells function form baseline to Month 12 (kinetics) | at Day1, Day2, Day9, Day30, Month3, Month6, Month12
  Immunomonitoring: NK ontogeny after in vivo transfer, characterization of KIR expression (phenotype and genotype), documentation of functional activity against tumor cell line and EBV transformed B cell lines. These studies will allow calibrating further the kinetics of NK cells function (cytotoxicity and cytokine production) as well to answer different questions of fundamental immunology
  The following studies will be performed:
  1. Analysis of early steps of aGVHD, immune activation and toxicity
  2. Impact of the infusions on NK reconstitution and myeloid cells including dendritic cells
  3. Antileukemic effects

CONTACTS AND LOCATIONS:
Overall Officials: BLAISE Didier, MD PhD, Principal Investigator — Institut Paoli-Calmettes
Locations (1):
- Institut Paoli-Calmettes, Marseille, France

REFERENCES:
- [Derived] Mfarrej B, Gaude J, Couquiaud J, Calmels B, Chabannon C, Lemarie C. Validation of a flow cytometry-based method to quantify viable lymphocyte subtypes in fresh and cryopreserved hematopoietic cellular products. Cytotherapy. 2021 Jan;23(1):77-87. doi: 10.1016/j.jcyt.2020.06.005. Epub 2020 Jul 25. PMID 32718876
- See also: official web site of the sponsor — http://www.institutpaolicalmettes.fr/